CLINICAL TRIAL: NCT06592651
Title: Home Within the Heart
Brief Title: Home Within the Heart: a Playful Journey to Strengthen Family Resilience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Yael Enav, Head of Emotiinal Regulation and Mentalization Lab, University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 003/24
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Family Resilience; Short-term Therapy; The Integration of Narrative Therapy and Play Therapy
Keywords: Play therapy; Family Resilience; Reflective function; Situational anxiety; Children's mental well-being; Parental mental well-being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parental Reflective Functioning intervention Group (Experimental): participants will attend four psycho-educational workshop sessions, where they will learn strategies for emotion regulation and mentalization to enhance open and secure communication within the family, strengthen the parent-child bond, and reinforce feelings of safety and stability.
  Interventions: Behavioral: Play Therapy Workshop

INTERVENTIONS:
Behavioral: Play Therapy Workshop — 4 session group intervention foucused on psycho-educational knowledge regarding tools for effective emotional coping with stressful events in the context of the "Iron Swords" war, focusing on building mental resilience in the parent-child dyad through play therapy. Each group consists of 5 parent-child dyads with children aged 3-6 years, who have been evacuated from war zones in the northern and southern regions of the country.

SUMMARY:
The primary aim of this clinical trial is to enhance open and secure communication within the family, strengthen the parent-child bond, and reinforce feelings of safety and stability, and strengthen family resilience.

In addition,the investigators want to assess the effectiveness of a short-term therapeutic workshop in enhancing reflective functioning, beliefs about the malleability of emotions, the reported use of effective emotional regulation strategies, and the perceived parental self-efficacy and child behavior.

DETAILED DESCRIPTION:
The participants will:

Complete questionnaires and participate in clinical interviews regarding their relationship with their children and their mental functioning prior to the workshop.

The intervention group will engage in a 4-session workshop (held once a week) facilitated practitioners from various therapeutic disciplines, including clinical, educational, and developmental psychologists, as well as group facilitators.

During each session, observers document the quality of the interaction between the parent and child, focusing on aspects such as emotion, responsiveness, encouragement, and instruction.

After the workshop, participants will again complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

A parent who have been evacuated from war zones in the northern and southern regions of the country, and has a child of ages 3-6.

Exclusion Criteria:

* A parent under the age of 18.
* A parent who have not been evacuated from war zones.
* A parent who has a child under 3 years of age, or above 6 years of age.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scales-21 (DASS-21) | Up to 20 weeks
  DASS-21 is a widely used psychological assessment tool designed to measure the emotional states of depression, anxiety, and stress.Each item is scored on a 4-point Likert scale ranging from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time"). The scores for each subscale are summed and then multiplied by 2 to maintain consistency with the original DASS-42 scores.

SECONDARY OUTCOMES:
Mental Health Continuum-Short Form (MHC-SF) | Up to 20 weeks
  The MHC-SF is a shorter version of the Mental Health Continuum-Long Form (MHC-LF) and is designed to assess well-being across three dimensions: emotional well-being, social well-being, and psychological well-being.Each item is rated on a 6-point Likert scale, ranging from 0 ("never") to 5 ("every day"). The responses reflect the frequency of these positive experiences over the past month. Scores are calculated for each dimension, and a total score is obtained by summing the items. Higher scores indicate higher levels of well-being.
Parental Reflective Functioning Questionnaire (PRFQ-18) | Up to 20 weeks
  The PRFQ-18 questionnaire consists of 18 items which respondents rate each item on a 7-point Likert scale, where higher scores indicate higher levels of reflective functioning.
Political Life Events Exposure (PLE) | Up to 20 weeks
  Political Life Events Exposure will be measured using the PLE scale containing 20 items regarding injury to a family member as a result of war, terrorism or military circumstances. For each item, participants are asked to indicate if they were exposed over the past six months, and if so, how stressful it was for them on a 5-point Likert scale from 1 (not at all) to 5 (very stressful) .Two measures are calculated: objective exposure (the sum of events that individuals experience) and subjective exposure (the sum of ratings of the stress level associated with the event). There is no justification for calculating an internal consistency score for PLE, but test-retest reliability has revealed a high reliability of r=0.87.
Stress Reaction Checklist (SRCL) | Up to 20 weeks
  The Stress Reaction Checklist (SRC) or Stress Reaction Checklist for Life Events (SRCL) is a psychological assessment tool designed to measure an individual's stress reactions following life events. This tool evaluates the cognitive, emotional, behavioral, and physical responses to stress, providing insights into how individuals cope with stressful situations.Responses are typically measured on a 5-point Likert scale,with higher scores indicating more severe or frequent stress reactions. The total score can be used to assess overall stress levels, while subscale scores can provide detailed information about specific types of stress responses.
Child-Parent Relationship Scale - Short Form (CPRS-SF) | Up to 20 weeks
  The Child-Parent Relationship Scale - Short Form (CPRS-SF) consists of 15 items designed to assess the quality of the parent-child relationship. These items are divided into two subscales: Closeness Subscale and Conflict Subscale. Respondents (typically parents) rate each item on a Likert scale, often ranging from 1 (definitely does not apply) to 5 (definitely applies).The scale provides scores for the overall relationship quality as well as specific subscales for warmth, closeness, and conflict.
Brief Parental Self-Efficacy Scale (BPSES) | Up to 20 weeks
  The BPSES typically consists of 6 to 10 items, although this can vary depending on the specific version used. Each item is rated on a 5-point Likert scale, often ranging from 1 (Strongly Disagree) to 5 (Strongly Agree), where parents indicate their level of agreement with statements about their parenting abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Mayer, Phd, Principal Investigator — University of Haifa; Yael Enav, Phd, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
All IPD excluding personal information given by participants in interview (records and transcripts), however coded information for these interview will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 2 years after publication of the primary study results and will be available for 5 years.
Access Criteria: Eligibility*: Access restricted to reseachers affiliated with accredited academic institutions or healthcare organizations with relevant credentials.
  Application*: Sumbit application form, research roposal, and CV to the principal investigator or designated contact.
  Review and Approval*: Applications reviewed by the data access committee. Decision within 4-6 weeks.
  Conditions of Use*: Data to be used solely for the approved project. Maintain confidentiality and data security. No third-party sharing withour approval.
  Publicatins and Reorting*: Sumbit summary or findings within 12 months.Acknowledge original study in publications and provide copies to the principal investigator.
URL: https://drive.google.com/drive/folders/1tf_1fbKCJjbqveJVIvTZ43_OdtA6aE-c